CLINICAL TRIAL: NCT02893618
Title: A 5 Treatment Period Crossover Pharmacokinetic Study Evaluating Dose Proportionality and Food Effects of Diazoxide Choline Controlled-Release Tablet (DCCR)
Brief Title: A 5 Treatment Period Pharmacokinetic Study Evaluating Dose Proportionality and Food Effects of Diazoxide Choline Controlled-Release Tablet (DCCR)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Essentialis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PK024
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- DCCR 75 mg fasted (Experimental): Administered a single 75 mg dose of DCCR after an overnight fast followed by 4 hours of fasting
  Interventions: Drug: Diazoxide choline controlled-release tablet
- DCCR 150 mg fasted (Experimental): Administered a single 150 mg dose of DCCR after an overnight fast followed by 4 hours of fasting
  Interventions: Drug: Diazoxide choline controlled-release tablet
- DCCR 300 mg fasted (Experimental): Administered a single 300 mg dose of DCCR after an overnight fast followed by 4 hours of fasting
  Interventions: Drug: Diazoxide choline controlled-release tablet
- DCCR 450 mg fasted (Experimental): Administered a single 450 mg dose of DCCR after an overnight fast followed by 4 hours of fasting
  Interventions: Drug: Diazoxide choline controlled-release tablet
- DCCR 300 mg fed (Experimental): Administered a single 300 mg dose of DCCR after a standardized meal
  Interventions: Drug: Diazoxide choline controlled-release tablet

INTERVENTIONS:
Drug: Diazoxide choline controlled-release tablet — QD tablet formulation of choline salt of diazoxide
  Other Names: DCCR

SUMMARY:
Open label, parallel-group, single site, 5 treatment-period study with 4 dose levels of DCCR, 1 of which is administered both with and without food.

DETAILED DESCRIPTION:
Open label, parallel-group, single site, 5 treatment-period study with 4 dose levels of DCCR, 1 of which is administered both with and without food, with a 10 Day washout period between treatments. There will be 8 treatment sequences with 4 subjects randomized to each.

ELIGIBILITY:
Inclusion Criteria:

* Ability to follow verbal and written instructions
* Informed consent form signed by the subject
* Completed screening within 7 days prior to dosing
* BMI between 18.5 and 35 kg/m2
* Generally healthy
* fasting glucose less than or equal to 100 mg/dL
* HbA1c less than or equal to 6%

Exclusion Criteria:

* Pregnancy or breast feeding
* absence of contraception
* administration of investigational drug within 1 month prior to screening
* anticipated requirement for prohibited medication (systemic corticosteroids or anti-diabetic medications)
* allergic reaction to or significant intolerance of diazoxide, thiazides or sulfonamides
* known type 1 or type 2 diabetes mellitus
* congestive heart failure
* gastric bypass surgery
* history of drug or alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-07; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters: Cmax | up to 24 hours
  Cmax derived from PK samples taken at 0, 1, 3, 6, 9, 12, 15, 18, 21 and 24 hours post-dose
Pharmacokinetic parameters: AUC0-24 | up to 24 hours
  AUC0-24 derived from PK samples taken at 0, 1, 3, 6, 9, 12, 15, 18, 21 and 24 hours

SECONDARY OUTCOMES:
Pharmacokinetic parameters: CL/F | up to 24 hours
  CL/F derived from PK samples taken at 0, 1, 3, 6, 9, 12, 15, 18, 21 and 24 hours
Pharmacokinetic parameters: Tmax | up to 24 hours
  Tmax derived from PK samples taken at 0, 1, 3, 6, 9, 12, 15, 18, 21 and 24 hours

IPD SHARING:
Plan to Share IPD: Undecided